CLINICAL TRIAL: NCT03789981
Title: Exploring Disease Immunogenicity and the Immunological Effects of Hypomethylating Agents in Acute Myeloid Leukemia
Acronym: Immune-AML
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRSTB082
Record Dates: First submitted 2018-11-08; First posted 2018-12-31 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; Immunogenic profile; transcriptome analysis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow (BM) and peripheral blood (PB) and saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- At diagnosis: Immunogenic profile in patients affected by primary or secondary AML at diagnosis
  Interventions: Genetic: Immunogenic profile
- At relapse: Immunogenic profile in patients affected by primary or secondary AML at relapse
  Interventions: Genetic: Immunogenic profile

INTERVENTIONS:
Genetic: Immunogenic profile — RNA sequencing (RNAseq), Whole exome sequencing (WES), NeoAntigens (NeoAg), Immune checkpoints analysis, Gene expression profiling

SUMMARY:
This is a multicenter, prospective, translational study, to evaluate the immunogenic profile of AML cases according to immune checkpoint molecule expression.

DETAILED DESCRIPTION:
This is a multicenter, prospective, translational study. Pharmacological treatments will not be object of the present study. Patients will follow the prescribed therapeutic indications according to regular clinical practice. Biological samples and clinical data will be collected at fixed timepoints.

Aim of the study is to evaluate the immunogenic profile of AML cases according to immune checkpoint molecule expression.

A total of 75 AML patients affected by primary or secondary AML, at diagnosis ( 45 patients) or relapse (30 patients) will be enrolled in the protocol (18 months for patient enrolment). Blood,BM and saliva samples will be collected from each patients; for patients enrolled at diagnosis, samples will be collected before and after treatment with hypomethylating agents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with new diagnosis of primary or secondary AML candidate to first line treatment with hypomethylating agents (specific for Cohort 1) Patients with primary or secondary AML who relapse after/during first line treatment with hypomethylating agents (specific for Cohort 2)

   for each cohort:
2. Participant is willing and able to give informed consent for participation in the study
3. Male or Female, aged >18 years
4. Availability of clinical data

Exclusion Criteria:

1. Age < 18 years
2. AML M3 subtype according to FAB classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AML patients affected by primary or secondary AML, at diagnosis or relapse
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Immunogenic profile of primary or secondary AML patients in according to the variations in expression of molecules involved in immune checkpoint | up to 30 months
  The immunogenic profile of AML cases obtained by NeoAgprediction will be related with established biological and clinical parameters (including karyotype, percentage of blasts, clinical outcome) performing RNA sequencing (RNAseq) and whole exome sequencing (WES) analysis

SECONDARY OUTCOMES:
Investigation of the relationship between leukemia immunogenicity and immune checkpoint activation | up to 30 months
  the relationship between leukemia immunogenicity and immune checkpoint activation through transcriptome analysis of downstream pathways by flow cytometric analysis
Investigation of the activation of immune checkpoint molecules | up to 30 months
  Investigation of the activation of immune checkpoint molecules under the selective pressure of hypomethylating agents treatment by gene expression profilling
The investigation of the association of the immune checkpoint status with clinical outcomes | up to 30 months
  Investigation of the association of the immune checkpoint status with clinical outcomes (OS, PFS) estimated according to Kaplan-Meier.
The investigation of the association of the immunogenic profile with clinical outcomes | up to 30 months
  Investigation of the association of the immunogenic profile with clinical outcomes (OS, PFS) estimated according to Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (14):
- Italy (14):
  - AO Spedali Civili di Brescia, Brescia, BS
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - IRCCS Casa sollievo sofferenza, San Giovanni Rotondo, FOGGIA
  - IRCCS AOU S. Martino Genova, Genova, GE
  - Ospedale G. Da Saliceto, Piacenza, PC
  - Irccs Crob, Rionero in Vulture, PZ
  - Osp. S. Maria delle Croci, Ravenna, RA
  - Ospedale degli Infermi, Rimini, RN
  - AOU Senese, Siena, SI
  - Università di Torino, Orbassano, TO
  - AO Ordine Mauriziano di Torino, Torino, TO
  - Azienda ULSS2 Marca Trevigiana, Treviso, TV
  - AOU Maggiore della Carità, Novara
  - AOU di Udine, Udine